CLINICAL TRIAL: NCT04438369
Title: Evaluation of Ultrasound-guided Erector Spinae Block for Postoperative Analgesia in Laprascopic Ventral Hernia Repair.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018/2239
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-04

CONDITIONS: Ventral Hernia; Postoperative Pain; Regional Anesthesia
Keywords: Erector Spinae Plane Block; Postoperative pain; Ventral hernia repair
MeSH Terms: conditions — Hernia, Ventral; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The study is planned as a randomized controlled trial (RCT) with two study arms. One arm is the intervention arm, who will receive the active treatment. The other arm is the control arm, who will receive a placebo treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization was done through a computer-generated block randomization process (randomization.com) to reduce bias. The block sizes were randomly chosen to 2, 4 and 6. The total patients randomized were 60 patients to account for missing data and protocol violations. A study nurse prepared and placed the notes of study allocation covered with aluminum foil into opaque envelopes. The envelopes were numbered from 1- 70.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae block (Active Comparator): Group ESPB: Multimodal analgesia comprising of preoperative paracetamol adjusted for weight (2000 milligrams (mg) >70 kilograms (kg) <70 years, 1500 mg <70 kg >70 years, 1000 mg <50 kg) and diclofenac adjusted for weight (100 mg >70 kg <70 years, 50 mg <70 kg >70 years). After the operation they receive paracetamol 1000 mg x4 and diclofenac 50 mg x3 a day, as well as PCA with iv oxycodon 1 mg/ml.
  Preoperatively positioned bilateral catheters at level T7 injected with ropivacaine 2,5 mg/ml, 30 ml on each side. Postoperative maintenance treatment with injection of 2 mg/ml ropivacaine 30 ml on each side every 6 hours postoperatively. Maximum allowed bolus preoperative ropivacaine dose is 3 mg/kg body weight (BW), while the maximum 24 hour dose postoperatively is 11 mg/kg to avoid local anesthesia systemic toxicity (LAST). The catheter will be discontinued 24 hours after the original procedure. The container with ropivacaine will be masked for blinding of the personnel on the ward.
  Interventions: Procedure: Erector Spinae Plane Block
- Control (Placebo Comparator): Control group with standard multimodal analgesia: Preoperative paracetamol adjusted for weight (2000 milligrams (mg) >70 kilograms (kg) <70 years, 1500 mg <70 kg >70 years, 1000 mg <50 kg) and diclofenac adjusted for weight (100 mg >70 kg <70 years, 50 mg <70 kg >70 years). After the operation they receive paracetamol 1000 mg x4 and diclofenac 50 mg x3 a day, as well as PCA with iv oxycodone 1 mg/ml.
  Insertion of bilateral catheters preoperatively. Injection of 30 ml saline preoperatively and every 6 hours postoperatively. The catheter will be discontinued 24 hours after the original procedure. The container with saline will be masked for blinding of the personnel on the ward.
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Cathether based Erector Spinae Plane Block for postoperative pain management.

SUMMARY:
Ventral hernia repair is associated with significant postoperative pain, and regional anesthetic techniques are of potential benefit.

The postoperative mobility and training is of utmost importance in this patient group, and could be increased using local anesthetics instead of opioids.

Inadequate post-operative pain control can lead to adverse consequences for patients, such as the development of chronic pain, immunosuppression, poorer healing of surgical wounds, as well as adrenergic activation and its consequences in the form of coronary incidents or gastrointestinal obstruction and postoperative nausea and vomiting (PONV). Moreover, lack of mobility can result in thrombosis and embolism. These complications affect hospital functioning, which leads to decreased patient satisfaction, a worse reputation for the hospital, longer stays in the recovery room, prolonged hospitalizations, higher incidence of re-surgeries and re-admissions, and higher costs for care and treatment.

Erector spinae plane block (ESPB) is the latest of the truncal blocks and was first described in 2016. The efficacy of bilateral ESPB at the T7 level has been described in a study of 4 cases, moreover effective analgesia with ESPB after bariatric surgery has been described in a study of 3 cases. When performed at the level of the T7 transverse process, studies show the potential to block both supra-umbilical and infra-umbilical dermatomes. So far there are mostly case studies done in this field of study, and internationally there is a call for research into the effect of this technique and randomized controlled trials.

The objective of this study is to compare ESPB to multimodal analgesia in patients undergoing ventral hernia repair.

DETAILED DESCRIPTION:
Hypothesis, aims and objectives

The postulated nullhypothesis and alternativ hypothesis is:

H0= there is no difference in opioid consumption postoperatively between multimodal analgesia and ESPB. HA= there is a reduction in opioid consumption postoperatively between standard multimodal analgesia and ESPB.

Sample size calculation

Sample size estimation was calculated from our series of 20 pilot-patients on ventral hernia surgery without block, who needed on average 24.6 mg oral morphine equivalents (OME) iv oxycodone rescue analgesia during the first hour, SD=17.35 mg. Assuming a one sided study and in order to show a 50% reduction in rescue opioid consumption after a successful block with 80% power and 0.05 as level of significance, at least 2 x 26 patients should be studied, total of 52 patients. In order to adjust for missing data and protocol violations we decided to include 2 x 30 patients in our study.

This is a study where all parties are blinded for the allocation. A study nurse draws up the allocated study medication in an unmarked syringe so that the anesthesiologist is blinded. The study nurse responsible for the medication is not the same nurse that does the postoperative scoring. The study nurse responsible for the medication puts masked containers of the allocated medication into opaque envelopes and delivers the envelope to the ward. The ward personnel will then be masked for the allocation. The study nurse responsible for the follow up calls are not the same study nurse responsible for the medications and as such is also blinded for the allocation.

The primary outcome measure is the opiate consumption measured in oral morphine equivalents after 1 hour.

Secondary outcome measures are;

* Opiate consummation after 4 hours, 24 hours, 48 hours and 7 days. As patients receive different types of opiates, opiate consumption will be measured as oral morphine equivalents for ease of comparison. Oksykodon iv is converted by a factor of 1:1,5 to oral morphine.
* Time to first mobilization
* Time to first analgesic requirement
* Pain measuring tool used in this project is the validated numerical rating scale (NRS), which is a 11- point scale from 0-10, where no pain is NRS=0, mild pain is NRS 1-3, moderate pain NRS 4-6 and severe pain 7-10. NRS will be measured at rest and with activity at the time points 1, 2 and 3 hours.
* Sedation is measured by the validated Pasero opioid-induced sedation scale (POSS). The POSS measures normal sleep as S and then the degree of sedation on a numerical scale from 1-4. Will be measured at 1, 2 and 3 hours.
* Nausea and vomiting is measured by the validated PONV impact scale. This is a tool that entails two questions about nausea and vomiting, and each question gets rated on a numeric scale from 0-4. Will be measured at 1, 2 and 3 hours.

After the operation the patients will be asked to answer the QoR-15, which consist of 15 questions distributed on two dimensions: "physical" and "mental" well-being, where the patients report their experiences on a scale from 0 (=not at all) to 10 (=all the time). As a complementing measure to the QoR-15 the patients will also be asked the EQ-5D questionnaire. The EQ-5D questionnaire is an outcome measure of patient health after operation. The EQ-5D-5L is comprised of two different measures; the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). Both QoR-15 and EQ-5D will be measured at 48 hours and 7 days.

The objective is to gain knowledge to support anesthesiologists when deciding analgesic approach, as well as in shared decision-making with patients (including the patient perspective). All results are expected to be presented during the project period.

ELIGIBILITY:
The inclusion criteria:

* Age >18
* BMI (body mass index) 18,5 - 40 and weight >65 kg
* ASA (American Association of Anesthesiologists Classification system for physical status) I-III .
* Scheduled for elective ventral hernia operation
* Planned hospital stay >24 hrs

The exclusion criteria;

* Allergy to latex, local anesthesia, Non-Steroidal Anti-Inflammatory Drugs or opioids
* Diabetes
* Chronic pain with daily opiate use
* Patients with severe renal and/or hepatic disease
* Local infection at the site of injection
* Systemic infection
* AV block 2-3
* Inability to understand written or spoken Norwegian
* Inability to cooperate
* Dementia
* Known abuse of alcohol or medication
* Pregnancy
* Weight under 65 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Opiat consumption | Postoperatively at one hour.
  The opioid consumption measured in orale morphine equivalents after one hour postoperatively.

SECONDARY OUTCOMES:
Postopertive nausea | Postoperatively at 0-4 hours, 4-24 hours, 24-48 hours and 48 hours-7 days.
  We will measure postoperative nausea with the Postoperative nausea and vomiting (PONV) impact scale. This is a tool that entails two questions about nausea and vomiting, and each question gets rated on a numeric scale from 0-4.
Postoperative sedation | Postoperatively at 0-4 hours, 4-24 hours, 24-48 hours and 48 hours-7 days.
  We will measure postoperative sedation with the Pasero opioid-induced sedation scale (POSS). The POSS measures normal sleep as S and then the degree of sedation on a numerical scale from 1-4. Will be measured at 1, 2 and 3 hours.
Postoperative pain | Postoperatively at 1-4 hours, 4-24 hours, 24-48 hours and 48 hours-7 days.
  We will measure postoperative pain with postoperative Numeric Rating Scale (NRS). A scale from 0-10 where 0 is no pain and 10 is worst pain imaginable.
Quality of recovery 15 | 24 hours, 48 hours and 7 days.
  We will measure the patients quality of recovery with the validated QoR-15 questionaire. This will be done via telephone interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Soerenstua, MD, Principal Investigator — Sykehuset Ostfold HF
Locations (1):
- Ostfold Hospital Trust, Moss, Moss, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At publication date and for three months.

REFERENCES:
- [Derived] Sorenstua M, Raeder J, Vamnes JS, Leonardsen AL. Evaluation of the Erector spinae plane block for postoperative analgesia in laparoscopic ventral hernia repair: a randomized placebo controlled trial. BMC Anesthesiol. 2024 May 29;24(1):192. doi: 10.1186/s12871-024-02566-x. PMID 38811911